CLINICAL TRIAL: NCT05085535
Title: Study of the Effect of Adding Manual Therapy to Therapeutic Exercise Programs in Older Adults With Limited Mobility and Pain Secondary to Aging.
Brief Title: Study of Manual Therapy Plus Therapeutic Exercise in Geriatrics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants were recruited for a quality study
Sponsor: Juan Vicente, López Díaz (Other)
Collaborators: Omphis Foundation (Other)
Responsible Party: Sponsor-Investigator, Juan Vicente, López Díaz, Director, Omphis Foundation
Organization: Omphis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TM-ET
Record Dates: First submitted 2021-09-21; First posted 2021-10-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain; Disability Physical; Aging Disorder
Keywords: Therapeutic exercise,; manual therapy,; elderly,; geriatrics,; pain,; disability.
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Intervention Model Description: It is a study of the randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A triple blinding will be carried out: 1) of the patient, 2) of the collaborator who performs the data collection, 3) of the computer data analyst.
  The physiotherapist who performs the intervention of manual therapy, exercise teaching and pain education, it is impossible to blind him.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): to which the treatment of therapeutic exercise and pain education will be applied,
  Interventions: Other: Exercise
- Manual Therapy (Experimental): to which the same treatment as the control group will be applied, adding manual therapy sessions based on musculoskeletal rhythmic mobilizations.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — Exercises for body mobility and muscle toning, Sophrology, musculoskeletal oscillatory manual therapy
  Arms: Manual Therapy
Other: Exercise — Exercises for body mobility and muscle toning, Sophrology
  Arms: Exercise

SUMMARY:
This research project is part of the process of generating scientific evidence, on whether the clinical results obtained, in the treatment of the consequences of aging on mobility, pain and disability, are better if therapeutic exercise programs are added sessions of manual therapy and training in pain awareness, or on the contrary, do not significantly modify the effect of exercise programs.

DETAILED DESCRIPTION:
General objective:

Find out if adding Manual Therapy (MT) sessions to therapeutic exercise programs increases the efficacy of clinical results for the treatment of ailments derived from aging in older adults (65 <age <85).

Specific objectives:

1. Assess the effects on pain. (hypothesis: MT improves pain outcomes)
2. Assess the effects on physical disability. (hypothesis: MT improves results regarding physical disability)
3. Assess the effects on mental disability. (hypothesis: MT improves results regarding mental disability)
4. Assess the effects on the prevention of falls (hypothesis: MT improves the results regarding the risk of falls)

Methodology:

Study design: It is a study of the randomized clinical trial type, with triple blind.

Selection of participants:

1. General criteria:

* The sample will be selected from the patients who volunteer to participate in the study, which will be announced by the media (Radio and / or TV) and meet the inclusion criteria and not the exclusion criteria.
* Participants will be treated by different therapists, who will be instructed in the treatments to be performed on the participants, to eliminate the therapist's personal factor as a contaminating variable.
* Participants will be referred to the physiotherapist according to the group assigned by the randomization process, which will be unknown by the patient.

Sample size:

To calculate the sample size, the EPIDAT 4.2 or GRANMO 7.12 computer program will be used, depending on the population and epidemiological data of the Catalunya area, of older adults, with disabilities and mechanical-degenerative pain.

If the calculation is made based on a Student's t test for independent data, accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 25 subjects would be required in each group to detect a minimum difference of 20 percentage points. between two groups, assuming a common standard deviation of 25 points, and a loss to follow-up rate of 0%, following the usual criteria of biostatistics in health sciences (1) and the criteria of minimal differences between groups previously used in similar pilot studies.

In case of loss of subjects in the sample, participants should be replaced by others to maintain proportions. The definitive calculations will be made with more precision after the epidemiological study mentioned above.

Randomization Of all the participants who meet the inclusion criteria and do not have any exclusion criteria, a number will be assigned, after being randomized through a computerized process, to distribute each number to the corresponding group. The patient will not know which group he has been assigned to.

Analytical procedure:

Analysis by computer processing with SPSS 22.0 ® program. Performed by a blinded computer analyst.

Ethical aspects:

During the study, national and international guidelines (code of ethics, Declaration of Helsinki) will be followed, as well as the legal regulations on data confidentiality (Organic Law 3/2018 of December 5 on the Protection of Personal Data and guarantee of digital rights -LOPD-).

ELIGIBILITY:
Inclusion Criteria:

* People of both sexes.
* Between 65 and 85 years of age.
* No acute pathologies at the time of selection.
* Who present symptoms of muscle-joint degenerative mechanical aging with an intensity score greater than 4 on a scale of 0-10.

Exclusion Criteria:

* Patients with a recent traumatic history.
* Presence of an acute-type radiation component of neurological origin to upper or lower limbs.
* With neurological alterations both central and peripheral.
* Who are taking opioid-based analgesic medication, gabapentin, etc.
* Patients with severe malformations.
* Who are following any other type of treatment, be it manual or physical agents or alternative or complementary therapies.
* Those who have been treated with infiltrations or the like in a period of less than a year before starting the study.
* Patients with a serious psychiatric history such as schizophrenia or psychopathies.
* Patients with cognitive impairment.
* Patients with vestibular problems that cannot tolerate oscillatory movements.
* Those who are contraindicated due to their general metabolic or cardiopulmonary state to carry out moderate physical exercise.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-08 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of subjective assessment of pain intensity | beginning and through study completion, an average of 12 weeks
  using a VAS TEST (Visual Analog Score for pain) (Minimum = 0 better and maximum = 10 worse)
Change of the qualitative aspects of pain | beginning and through study completion, an average of 12 weeks
  using the McGill pain questionnary
Change of of disability and health status | beginning and through study completion, an average of 12 weeks
  using the SF36 test (36-item short form health survey)

SECONDARY OUTCOMES:
Change of risk of falls | beginning and through study completion, an average of 12 weeks
  Tinetti test. (test for balance and gait) (Minimum = 0 worse and maximum = 28 better)
Change of Physical activity in older adults | beginning and through study completion, an average of 12 weeks
  PASE test (Physical Activity Scale for the Elderly)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Vicente López Díaz, Principal Investigator — Fundación Omphis

IPD SHARING:
Plan to Share IPD: No